CLINICAL TRIAL: NCT03978975
Title: Effect of Water Temperature on Energy Response During Aquatic Cycling in Women: Impact of Weight Status
Brief Title: Water Exercise and Health (WATHEALTH)
Acronym: WATHEALTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: SSR Obésité Nutrition UGECAM (Unknown); Aquafit Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2018 DUCLOS 4 (Wathealth); 2019-A00353-54 (Other: ANSM)
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Overweight; Hunger
Keywords: Energy expenditure; Food intake; Women; aquacycling
MeSH Terms: conditions — Overweight | interventions — Eating

STUDY DESIGN:
Intervention Model Description: participants may receive different interventions sequentially during the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal weight women (Active Comparator): 20 women with a body mass index ranging between 18,5 and 24,9 kg.m2
  Interventions: Behavioral: Food intake
- overweight women (Experimental): 20 women with a body mass index ranging between 25 and 29,9 kg.m2
  Interventions: Behavioral: Food intake

INTERVENTIONS:
Behavioral: Food intake — For all those session, subjects will take a standardized breakfast (570kcal) three hours before experimental session.
  Control session (CON): subject will stand sited without any activity during 40 min.
  Subjects will be submitted to three aquatic cycling exercise session:
  * session 27°C :aquatic cycling at 27°C without water jet during 40 min
  * session 27°C+ water jets : aquatic cycling at 27 °C with water jets during 40 min
  * session 18°C : aquatic cycling at 187°C without water jet during 40 min Every exercise session will be set at 70% of theorical maximal heart rate During each session, oxygen consumption and carbon dioxide production will be analysed with gas analysis system. Appetite and hunger sensation will be measured with a specific scale at different time point of each day of experimental session. Thirty minutes after the end of each experimental session subjects will have a buffet meal for lunch time.

SUMMARY:
Aquatic cycling is becoming more popular as it appears to be more suitable for men and women even with poor physical activity level. Commercial tagline highlight beneficial effect of this activity on weight management. However there are poor information concerning the energy response induced by this activity. The aim of this project is to investigate effect of water temperature on energetic response (energy expenditure and food intake) of cycling exercise in water in normal weight and overweight premenopausal women.

DETAILED DESCRIPTION:
After inclusion visit, all subject will be submitted to DXA to obtain body composition data. Then subjects will be submitted to four experimental session in a semi-randomized order. For all those session, subjects will take a standardized breakfast (570kcal) three hours before experimental session.

Control session (CON): subject will stand sited without any activity during 40 min.

Subjects will be submitted to three aquatic cycling exercise session:

* session 27°C :aquatic cycling at 27°C without water jet during 40 min
* session 27°C+ water jets : aquatic cycling at 27 °C with water jets during 40 min
* session 18°C : aquatic cycling at 187°C without water jet during 40 min Every exercise session will be set at 70% of theorical maximal heart rate During each session, oxygen consumption and carbon dioxide production will be analysed with gas analysis system. Appetite and hunger sensation will be measured with a specific scale at different time point of each day of experimental session. Thirty minutes after the end of each experimental session subjects will have a buffet meal for lunch time.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 40 years
* BMI under 25kg.m2 for normal weight women and between 25 and 29,9 kg.m2 for overweight women
* Daily breakfast
* Subject which approved informed consent
* Subject with French medical affiliation

Exclusion Criteria:

* Specific medical treatment
* Aquaphobia
* Subject under specific diet regimen or weight loss program
* Subject with cardio-vascular disease
* Surgical intervention less than 3 months
* Subject refusing informed and written consent
* Subject without French medical affiliation
* subject refusing inscription to the national voluntary list
* subject being in an exclusion period
* subject smoking or drinking alcohol frequently
* subject with intense physical activity

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-12-19 (Estimated); Study Completion 2022-01-19 (Estimated)

PRIMARY OUTCOMES:
Food intake during buffet meal 30 minutes after the end of experimental session | Day 7
  total energy intake at the post session lunch will be calculated by measuring food intake
Food intake during buffet meal 30 minutes after the end of experimental session | Day 14
  total energy intake at the post session lunch will be calculated by measuring food intake
Food intake during buffet meal 30 minutes after the end of experimental session | Day 21
  total energy intake at the post session lunch will be calculated by measuring food intake
Food intake during buffet meal 30 minutes after the end of experimental session | Day 28
  total energy intake at the post session lunch will be calculated by measuring food intake

SECONDARY OUTCOMES:
Appetite, hunger and satiety | Day 7
  using a visual analog scale from 0 millimeter (no sensation) to 100mm (highest sensation)
Appetite, hunger and satiety | Day 14
  using a visual analog scale from 0 millimeter (no sensation) to 100mm (highest sensation)
Appetite, hunger and satiety | Day 21
  using a visual analog scale from 0 millimeter (no sensation) to 100mm (highest sensation)
Appetite, hunger and satiety | Day 28
  using a visual analog scale from 0 millimeter (no sensation) to 100mm (highest sensation)
Energy expenditure | Day 7
  with a gas analyser energy expenditure will be measured in kcal
Energy expenditure | Day 14
  with a gas analyser energy expenditure will be measured in kcal
Energy expenditure | Day 21
  with a gas analyser energy expenditure will be measured in kcal
Energy expenditure | Day 28
  with a gas analyser energy expenditure will be measured in kcal
Perceived exertion | Day 7
  using Borg scale perceived exertion will be evaluated between 6 (very light) and 20 (extremely difficult)
Perceived exertion | Day 14
  using Borg scale perceived exertion will be evaluated between 6 (very light) and 20 (extremely difficult)
Perceived exertion | Day 21
  using Borg scale perceived exertion will be evaluated between 6 (very light) and 20 (extremely difficult)
Perceived exertion | Day 28
  using Borg scale perceived exertion will be evaluated between 6 (very light) and 20 (extremely difficult)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France